CLINICAL TRIAL: NCT02889653
Title: The Bleeding With Antithrombotic Therapy Study 2
Acronym: BAT2
Status: Completed | Type: Observational
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Kazunori Toyoda, Director and Chair, Department of Stroke and Cerebrovascular Diseases, National Cerebral and Cardiovascular Center, Japan
Other Study IDs: 16ek0210055h; 000023669 (Other: UMIN Clinical Trials Registry)
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Cerebrovascular and Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Any oral antithrombotics (antiplatelets or anticoagulants)

SUMMARY:
The purpose of this study is to determine the incidence and severity of bleeding complications in patients with cerebrovascular and cardiovascular diseases treated with oral antithrombotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cerebrovascular or cardiovascular diseases who start or continue taking oral antithrombotics (antiplatelets and/or anticoagulants) to prevent vascular events
* Patients who are able to receive MRI
* Provision of written informed consent either directly or by a suitable surrogate

Exclusion Criteria:

* MRI contraindication
* Any condition that in the opinion of the responsible physician or investigator that renders the patient unsuitable for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebrovascular or cardiovascular diseases who start or continue taking oral antithrombotics (antiplatelets and/or anticoagulants) to prevent vascular events in participating centers
Sampling Method: Non-Probability Sample
Enrollment: 5306 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
ISTH major bleeding | within 2 years

SECONDARY OUTCOMES:
Clinically relevant non-major bleeding | within 2 years
Hemorrhagic event details | within 2 years
Ischemic events and those details | within 2 years

CONTACTS AND LOCATIONS:
Locations (9):
- Japan (9):
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - St. Marianna University, Kawasaki
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Saga University, Saga
  - Tokushima University, Tokushima
  - Juntendo University, Tokyo
  - Kyorin University, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Koga M, Yoshimura S, Hasegawa Y, Shibuya S, Ito Y, Matsuoka H, Takamatsu K, Nishiyama K, Todo K, Kimura K, Furui E, Terasaki T, Shiokawa Y, Kamiyama K, Takizawa S, Okuda S, Okada Y, Kameda T, Nagakane Y, Yagita Y, Kario K, Shiozawa M, Sato S, Yamagami H, Arihiro S, Toyoda K; SAMURAI Study Investigators. Higher Risk of Ischemic Events in Secondary Prevention for Patients With Persistent Than Those With Paroxysmal Atrial Fibrillation. Stroke. 2016 Oct;47(10):2582-8. doi: 10.1161/STROKEAHA.116.013746. Epub 2016 Aug 16. PMID 27531346
- [Result] Takagi M, Tanaka K, Miwa K, Sasaki M, Koga M, Hirano T, Kamiyama K, Yagita Y, Nagakane Y, Hoshino H, Terasaki T, Yakushiji Y, Kudo K, Ihara M, Yoshimura S, Yamaguchi Y, Shiozawa M, Toyoda K; for BAT2 Investigators. The bleeding with antithrombotic therapy study 2: Rationale, design, and baseline characteristics of the participants. Eur Stroke J. 2020 Dec;5(4):423-431. doi: 10.1177/2396987320960618. Epub 2020 Sep 24. PMID 33598561
- [Result] Tanaka K, Miwa K, Takagi M, Sasaki M, Yakushiji Y, Kudo K, Shiozawa M, Tanaka J, Nishihara M, Yamaguchi Y, Fujita K, Honda Y, Kawano H, Ide T, Yoshimura S, Koga M, Hirano T, Toyoda K. Increased Cerebral Small Vessel Disease Burden With Renal Dysfunction and Albuminuria in Patients Taking Antithrombotic Agents: The Bleeding With Antithrombotic Therapy 2. J Am Heart Assoc. 2022 Mar 15;11(6):e024749. doi: 10.1161/JAHA.121.024749. Epub 2022 Mar 5. PMID 35253443
- [Derived] Miwa K, Tanaka K, Koga M, Tanaka K, Yakushiji Y, Sasaki M, Kudo K, Shiozawa M, Yoshimura S, Ihara M, Fujimoto S, Hoshino H, Kamiyama K, Kawano H, Nagasawa H, Nagakane Y, Nishiyama K, Yagita Y, Yoshimura S, Hirano T, Toyoda K; BAT2 Investigators. Prediction Model to Optimize Long-Term Antithrombotic Therapy Using Covert Vascular Brain Injury and Clinical Features. Stroke. 2025 Sep;56(9):2605-2616. doi: 10.1161/STROKEAHA.125.050859. Epub 2025 Jun 19. PMID 40534562